CLINICAL TRIAL: NCT01366482
Title: Directional AthErectomy Followed by a PaclItaxel-Coated BallooN to InhibiT RestenosIs and Maintain Vessel PatEncy: A Pilot Study of Anti-Restenosis Treatment
Brief Title: Atherectomy Followed by a Drug Coated Balloon to Treat Peripheral Arterial Disease
Acronym: DEFINITIVE AR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Collaborators: MEDRAD, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-4941
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Peripheral Arterial Disease; Claudication
Keywords: Peripheral arterial disease,; claudication,; atherectomy,; plaque excision,; drug-coated balloon; drug-eluting balloon
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Drug-eluting balloon (Experimental): Subjects are randomized to have a lesion treated with a paclitaxel-coated balloon Intervention: Cotavance Drug-Eluting Balloon
  Interventions: Device: Cotavance Drug-Eluting Balloon
- Plaque excision + drug-eluting balloon (Experimental): Subjects are randomized to have a lesion treated with plaque excision (PE) followed by treatment with a paclitaxel-coated balloon Intervention: SilverHawk/TurboHawk + Cotavance Drug-Eluting Balloon
  Interventions: Device: TurboHawk/SilverHawk + Cotavance Drug-Eluting Balloon
- Severely Ca++ Group (Experimental): Subjects with a severely calcified lesion will be assigned to a non-randomized arm and treated with plaque excision followed by a drug-eluting balloon Intervention: SilverHawk/TurboHawk + Cotavance Drug-Eluting Balloon
  Interventions: Device: TurboHawk/SilverHawk + Cotavance Drug-Eluting Balloon

INTERVENTIONS:
Device: Cotavance Drug-Eluting Balloon — Treatment with a paclitaxel-coated angioplasty balloon (without preceding plaque excision)
  Arms: Drug-eluting balloon
Device: TurboHawk/SilverHawk + Cotavance Drug-Eluting Balloon — Plaque excision with a SilverHawk or TurboHawk plaque excision device followed by treatment with a paclitaxel-coated angioplasty balloon
  Arms: Plaque excision + drug-eluting balloon
Device: TurboHawk/SilverHawk + Cotavance Drug-Eluting Balloon — Plaque excision followed by treatment with a paclitaxel-coated angioplasty balloon
  Arms: Severely Ca++ Group

SUMMARY:
The DEFINITIVE AR study is a prospective, multi-center, randomized pilot study evaluating the use of either the TurboHawk™ or SilverHawk® plaque excision systems followed by treatment with the Cotavance™ drug-eluting balloon catheter versus the Cotavance balloon catheter alone in patients with peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford Clinical Category 2-4
* At least 18 years of age
* Is able and willing to provide written informed consent prior to study specific procedures

Exclusion Criteria:

* Has a life expectancy of less than 24 months
* Is pregnant, of childbearing potential not taking adequate contraceptive measures, or nursing
* Has one or more of the contraindications listed in the SilverHawk/ TurboHawk or Cotavance IFUs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Target Lesion Percent Stenosis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Professor Thomas Zeller, Principal Investigator — Herz-Zentrum Bad Krozingen Germany; Professor Gunnar Tepe, Principal Investigator — Klinikum Rosenheim Germany
Locations (1):
- Imelda Hospital, Bonheiden, Belgium

REFERENCES:
- [Derived] Zeller T, Langhoff R, Rocha-Singh KJ, Jaff MR, Blessing E, Amann-Vesti B, Krzanowski M, Peeters P, Scheinert D, Torsello G, Sixt S, Tepe G; DEFINITIVE AR Investigators. Directional Atherectomy Followed by a Paclitaxel-Coated Balloon to Inhibit Restenosis and Maintain Vessel Patency: Twelve-Month Results of the DEFINITIVE AR Study. Circ Cardiovasc Interv. 2017 Sep;10(9):e004848. doi: 10.1161/CIRCINTERVENTIONS.116.004848. PMID 28916599